CLINICAL TRIAL: NCT04951401
Title: Pattern of Dyslipidemia Among Patients With Acute Coronary Syndrome at Sohag University Hospital
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Mostafa Abdelfattah, principal investigator, Sohag University
Other Study IDs: soh-Med-21-06-06
Record Dates: First submitted 2021-06-18; First posted 2021-07-06 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal & abnormal lipid parameters value: parameters value among normal and abnormal lipid profile
  Interventions: Other: lipid profile; Other: ECG

INTERVENTIONS:
Other: lipid profile — lipid profile
Other: ECG — ECG

SUMMARY:
In this study, I am aime to analyze lipid profile in patients with ACS who presents at sohag university hospital, and its clinical and complications pattern.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most important cause of death in men and women The great majority of ACS patients have at least one major risk factor.

Acute Coronary Syndrome (ACS) is a major reason for Coronary Care Unit ( CCU )sohag university hospital admission The risk of CAD was about 4 and 3 times higher in male and female smokers than nonsmokers respectively (Baba S et. al ; 2006) Dyslipidemia has been identified as one of most important modifiable risk factor for CAD . Treating dyslipidemia has clear benefits in the primary and secondary prevention of coronary heart disease (CHD) in both sexes . This study focused on dyslipidemia as a risk factor of acute coronary syndrome (ACS).

ELIGIBILITY:
Inclusion Criteria::

clinical diagnosed Acute coronary syndromes

-

Exclusion Criteria:

* chronic coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: about 100 adult patients will be included in this study aged above 18 years old diagnosed acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
dyslipiemia in acute coronary syndrome | one year
  pattern of dyslipidemia among patients with acute coronary syndrome at sohag university hospital

CONTACTS AND LOCATIONS:
Overall Officials: esraa m abdelfatah, resident, Principal Investigator — esraa m abdelfatah
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
dyslipidemia at acute coronary syndrome

REFERENCES:
- [Background] Graichen C, Tanner C. Diagnosis of Acute Coronary Syndrome. Am Fam Physician. 2018 Aug 1;98(3):Online. No abstract available. PMID 30215890
- [Background] Dali B. Clinical Profile, Dyslipidemia and ACS - a Correlation. JNMA J Nepal Med Assoc. 2014 Jul-Sep;52(195):907-13. PMID 26982665
- [Result] Ray KK, Ditmarsch M, Kallend D, Niesor EJ, Suchankova G, Upmanyu R, Anzures-Cabrera J, Lehnert V, Pauly-Evers M, Holme I, Stasek J, van Hessen MW, Jones P; dal-ACUTE Investigators. The effect of cholesteryl ester transfer protein inhibition on lipids, lipoproteins, and markers of HDL function after an acute coronary syndrome: the dal-ACUTE randomized trial. Eur Heart J. 2014 Jul 14;35(27):1792-800. doi: 10.1093/eurheartj/ehu105. Epub 2014 Mar 17. PMID 24639426
- [Result] Eisen A, Giugliano RP, Braunwald E. Updates on Acute Coronary Syndrome: A Review. JAMA Cardiol. 2016 Sep 1;1(6):718-30. doi: 10.1001/jamacardio.2016.2049. PMID 27438381